CLINICAL TRIAL: NCT01689883
Title: Improving Recovery After Stroke Via Electrical Stimulation of Proprioceptors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Wyss Institute at Harvard University (Other); Center for Integration of Medicine & Innovative Technology (Other)
Responsible Party: Principal Investigator, Yong-Tae Lee, Physiatrist, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-P-001592
Record Dates: First submitted 2012-09-10; First posted 2012-09-21 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Chronic Stroke Survivors
Keywords: stroke; electrical stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The investigators will use a system to inject small currents in the arm while subjects perform upper-limb movements. Subjects will perform multiple trials. During half of the trials, subjects will receive actual stimulation. During the other half, subjects will receive sham stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Current stimulator (Other): The investigators have developed a device to deliver very small currents to the arm. The device will be used while subjects perform upper-limb movements using a device for upper-limb rehabilitation. Subjects will perform multiple trials of movement. During half of the trials, they will receive actual stimulation. During the other half, they will receive sham stimulation.
  Interventions: Device: Current stimulator

INTERVENTIONS:
Device: Current stimulator — This is a device developed by the investigators to produce sub-sensory electrical stimulation delivered via subcutaneous electrodes placed on the skin.

SUMMARY:
The overall objective of the study is to test whether the use of small electrical currents to stimulate proprioceptors of the upper limb has potential for improving robot-assisted upper-limb rehabilitation in stroke survivors.

DETAILED DESCRIPTION:
Study participants will be instructed to perform upper-limb movements using a system designed for upper-limb rehabilitation (Armeo Spring by Hocoma AG). The system provides subjects with unloading of the stroke-affected arm thus facilitating the performance of upper-limb movements. The system will be used to track the movements of the stroke-affected arm. Simultaneously, a custom-designed system (a prototype developed by the investigators) will be used to deliver small electrical currents to the arm. We hypothesize that the currents delivered to the arm will improve the accuracy of the movements performed by study participants.

To assess if delivering small currents to the arm has an effect on the accuracy of the movements performed by the study participants, they will receive actual stimulation for some trials and sham stimulation for other trials. Because the investigators will deliver very small currents, study participants will be unable to perceive such currents and hence tell if they are performing the movements while receiving actual or sham stimulation. By comparing trials performed while subjects receive actual stimulation with trials performed while subjects received sham stimulation, the investigators will determine if the stimulation has an effect on the accuracy of the movements performed by the subjects.

It is worth noticing that the investigators collected primary outcome data to assess changes associated with the use of actual stimulation vs sham stimulation. Data during a follow-up session was also collected, but not for the purpose of collecting outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* unilateral and cortical, subcortical, or cerebellar stroke
* 6 months post-stroke
* Upper extremity impairments but able to move upper extremity against gravity 25% of the range
* Ability to understand directions and follow simple instructions
* Medically stable
* Upper Extremity Fugl-Meyer between 28 and 55
* At least four (4) months since last botox treatment
* Mini-Mental State Examination (MMSE) ≥ 23

Exclusion Criteria:

* Participation in other forms of therapy/ intervention for upper extremity motor recovery
* Upper extremity or trunk fractures
* Severe fixed contractures affecting the upper limbs
* Severe perceptual deficits or visual field impairments
* Severe cognitive deficits
* Pregnant women
* Presence of an implanted electrically operated medical device
* Evidence of more than one clinical stroke
* Serious medical or neurological illness
* History of head trauma or cerebral infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | Changes in Fugl-Meyer Assessment score with vs without stimulation
  Subjects are asked to perform upper-limb movements from which a therapist can assess the severity of movement abnormalities (e.g. flexion synergies)

SECONDARY OUTCOMES:
Jebsen-Taylor Hand Function Test | Changes in Jebsen-Taylor Hand Function Test score with vs without stimulation
  Subjects are asked to perform a set of functional movements from which a therapist can assess subjects' functional limitations
Motor Activity Log | Change in Motor Activity Log score with vs without stimulation
  Subjects are asked about the amount and quality of use of their stroke-affected arm during the performance of daily activities
Modified Ashworth Scale | Change in Modified Ashworth Scale score with vs without stimulation
  A therapist examines subjects to assess the severity of spasticity
Box and Block test | Change in Box and Block test score with vs without stimulation
  Subjects are asked to move as many small wooden blocks as possible from one to box to another in a set amount of time
Grip strength | Change in grip strength with vs without stimulation
  A hand dynamometer is used to measure grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No